CLINICAL TRIAL: NCT03336372
Title: Picato for the Treatment of Molluscum Contagiosum in Immunocompromised Patients
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor discontinued study on 8Sep2018
Sponsor: Center for Clinical Studies, Texas (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-Picato-1386
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — 3-ingenyl angelate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Picato topical gel (Experimental)
  Interventions: Drug: Picato

INTERVENTIONS:
Drug: Picato — Picato 0.05% or 0.015% topical gel applied nightly for 3 consecutive nights

SUMMARY:
Patients at least 18 years of age will be enrolled in the study to assess the efficacy and tolerability of Picato gel in the treatment of molluscum contagiosum. Patients must have an immunocompromised condition due to taking immunosuppressive drugs or having an inherited disease affecting the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female at least 18 years of age.
* Subject must have an immunocompromised condition due to use of immunosuppressive therapies for cancer or autoimmune disease treatment or prevention of organ transplant rejection or due to an inherited condition that affects the immune system.
* Subject has at least 10 clinically typical, visible and discrete MCs within a treatment area on either the face and/or trunk. Treatment area is defined as either:

  * One contiguous treatment area of at most 100 cm2
  * Two non-contiguous treatment areas totaling at most 100 cm2
* Subject must be willing to forego any other treatments of MC on the face and/or trunk, including tanning bed use and excessive sun exposure, throughout the duration of the trial.
* Subject is willing and able to participate in the study as an outpatient, making frequent visits to the study center during the treatment and follow-up periods, and to comply with all study requirements.
* Female subjects of childbearing potential must have a negative urine pregnancy test prior to trial treatment.
* Female subjects of childbearing potential must be willing to use effective contraception at trial entry and until the last follow-up visit at Week 24.

Exclusion Criteria:

* Location of the treatment area

  * on the periorbital skin
  * within 5 cm of an incompletely healed wound
  * within 10 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
* Previous participation in an ingenol mebutate trial.
* Treatment with ingenol mebutate gel in the treatment area within 6 months or outside of the treatment area within 30 days prior to study treatment initiation.
* Receipt of the following within 90 days prior to study treatment initiation:

  * interferons or interferon inducers
  * any dermatologic procedures or surgeries within the treatment area
* Receipt of any topical prescription medications in the treatment area within 30 days prior to study treatment initiation.
* Lesions in the treatment area have atypical clinical appearance (e.g. giant lesions greater than 5 mm, eczematous lesions, or folliculocentric lesions).
* Active dermatologic conditions that may confound the diagnosis of MC or would interfere with assessment of treatment, such as scabies, cutaneous lymphoma, or psoriasis.
* Clinical diagnosis/history or evidence of any medical condition that would expose a subject to an undue risk of a severe AE or interfere with assessments of safety and efficacy during the course of the trial, as determined by the (sub)investigator's clinical judgment.
* Known history of infection with Human Immunodeficiency Virus (HIV).
* History of melanoma.
* History of chronic alcohol or drug abuse within 12 months prior to screening, or any condition associated with poor compliance as judged by the (sub)investigator.
* Known or suspected allergy or reaction to any component of the IMP formulation.
* Patients who have experienced a clinically important medical event within 90 days prior to study treatment initiation (e.g., stroke, myocardial infarction, etc).
* Pregnant, breastfeeding, or lactating women.
* Participation in any another interventional clinical trial within 30 days prior to study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Complete clearance at Week 4 | 4 weeks
  Complete clearance is defined as no clinically visible MCs in the treatment area/

SECONDARY OUTCOMES:
Partial clearance at Week 4 | 4 weeks
  Partial clearance defined as at least 50% reduction in the number of clinically visible MCs in the treatment area.
Percentage of subjects who sustain complete clearance of MCs in the treatment area at Week 24 | 24 weeks
Percentage of subjects who clear MCs outside of the treatment area at Week 24 | 24 weeks

OTHER OUTCOMES:
Treatment Satisfaction Questionnaire for Medication | 24 weeks
  Scale range from "extremely satisfied" to "extremely dissatisfied".
EQ-5D-5L Index and Health Status | 24 weeks
  Scale range from 0 (worst health) to 100 (best health).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K Tyring, MD, PhD, Study Director — Center for Clinical Studies
Locations (1):
- Center for Clinical Studies, Houston, Texas, United States

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/72/NCT03336372/Prot_002.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT03336372/ICF_001.pdf